CLINICAL TRIAL: NCT07251985
Title: Cognitive Effects of Bioavailable Curcumin
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine and Chief of the Division of Clinical Nutrition at the University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25-1154
Record Dates: First submitted 2025-11-13; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Memory; Cognitive Function Decline
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theracurmin Super TS-P1 capsules containing 75 mg in total of curcumin will be administered orally) (Active Comparator)
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Theracurmin Super TS-P1 capsules containing 75 mg in total of curcumin will be administered orally (swallowed with water) twice a day (during breakfast and dinner) for 12 months
  Arms: Theracurmin Super TS-P1 capsules containing 75 mg in total of curcumin will be administered orally)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
An estimated 50% of older adults complain of memory changes that worsen as they age. Although numerous commercially available dietary supplements claim cognitive benefits, relatively few well-designed, longitudinal, placebo-controlled studies have rigorously evaluated their effects on cognitive performance.

In a previous double-blind, randomized, placebo-controlled, 18-month clinical trial in middle-aged and older non-demented adults, the investigators found that a bioavailable form of curcumin taken orally twice a day showed greater gains on specific measures of memory and attention relative to placebo. Although the investigators found significant between-group curcumin/placebo differences with moderate effect sizes, the sample size (n=40) was small. The present adequately powered, randomized, double-blind, placebo-controlled study will evaluate the effect of daily consumption of bioavailable curcumin on measurable changes in cognitive performance in non-demented middle-aged and older adults.

ELIGIBILITY:
Inclusion Criteria

1. Presence of age-related memory complaints;
2. Male or female aged 50 to 85 years of age at Visit 1.
3. performance on MoCA test of >= 18 (Milani et al, 2018)
4. Ability to perform normal daily activities independently (which excludes a diagnosis of dementia).
5. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
6. Agreement to participate in the entire study, which could last either 6 or 12 months depending on results of the interim analysis.
7. Adequate visual and auditory acuity for cognitive testing.
8. Screening laboratory tests that do not show significant medical problems that might interfere with study participation or impact cognitive test results.
9. Psychotropic medication, if used, should be stable for at least 2 weeks prior to randomization.
10. Agreement to avoid taking any curcumin, turmeric supplements or cognitive enhancing medicines or supplements during the course of the study.

Exclusion Criteria

1. Allergy to curcumin
2. Presence of a condition or abnormality that in the opinion of the site Principal Investigator would compromise the safety of the patient or the quality of the data.
3. Significant cerebrovascular disease or Alzheimer disease or any other dementia.
4. Neurological or physical illnesses that can produce cognitive deterioration.
5. History of myocardial infarction within the previous year or unstable cardiac disease.
6. Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100); significant liver or pulmonary disease, or cancer;
7. Current diagnosis of any major psychiatric disorder according to the DSM-IV TR criteria with a change in medication or clinical symptoms with the last 3 months prior to screening (APA, 2000).
8. History of alcoholism or substance addiction in the last 15 years.
9. Current treatment for seizure disorder;
10. Abnormal laboratory values with clinical significance in the opinion of the site Principal Investigator.
11. Current unstable medical illness including delirium, worsening congestive heart failure, unstable angina, recent myocardial infarctions, acute infectious disease, severe renal or hepatic failure, severe respiratory disease, metastatic cancer, or other conditions that, in the Principal Investigator's opinion, could interfere with the analysis of safety and efficacy in this study.
12. A 2-week washout is required prior to baseline for any of the following: curcumin or turmeric supplements, any anti-inflammatory medication other than occasional use (e.g., once per week).
13. The subject may not be an immediate family member (e.g., spouse, parent, child, sibling) of personnel directly affiliated with this study, the study site or study funding agency.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Memory | 12 months
  The primary endpoint will be a memory domain score calculated from the Consistent Long Term Recall score of the Buschke Selective Reminding Test (SRT)
Memory | 12 months
  Delayed Recall score of the Brief Visual Memory Test-Revised (BVMT-R).

SECONDARY OUTCOMES:
Cognitive function test | 12 months
  NIH TOOLBOX computerized set of cognitive tests
PROMIS Cognitive Function | 12 months
  Short Form 20a is a standardized questionnaire designed to assess an individual's self-reported cognitive abilities and problems over the past 7 days. It includes 20 items and is part of the Patient-Reported Outcomes Measure. The instrument produces a T-score standardized to the PROMIS metric. T-scores typically range from 20 to 80, with a population mean of 50 and standard deviation of 10.
Self-reported depression symptoms | 12 months
  Measured by Beck Depression Inventory (BDI). A 21-item self-report questionnaire assessing the severity of depressive symptoms. Total scores range from 0 to 63, with higher scores indicating more severe depression (i.e., a worse outcome).
Blood levels of curcumin | 12 months
  (to ensure adherence to protocol)
Inflammation and neurodegenerative markers | 12 months
  such as, TNF-α, C-reactive protein
metabolic markers | 12 months
  such as fasting glucose, insulin, C-peptide, glucagon, glucose-dependent-insulinotropic-polypeptide (GIP), HbA1C, and HOMA-IR index and lipid markers
Quality of life | 12 months
  Quality of life, SF-36: The SF-36 is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being. It measures each of the following eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health (about 15 minutes).
Body composition | 12 months
  Body composition will be assessed using an InBody bioelectrical impedance analysis (BIA) device.
APOE-4 carrier status | 12 months
  APOE-4 carrier status will be determined through genetic testing to identify whether participants possess at least one copy of the APOE 4 allele, a genetic risk factor associated with Alzheimer's disease.
Sleep quality | 12 months
  Pittsburgh Sleep Quality Index: PSQI will be employed to assess sleep quality. The PSQI is a widely recognized self-report questionnaire that evaluates sleep quality over a one-month interval. The PSQI comprises 19 self-rated items and an additional 5 items rated by bed partners or roommates. The self-rated items are used to calculate the total score, which ranges from 0 to 21. Each item on the PSQI is scored on a scale of 0 to 3, with 3 reflecting the highest level of dysfunction or disturbance. The scores of these items are then summed to compute a global PSQI score. A global PSQI score greater than 5 suggests significant sleep difficulties. A higher total score is indicative of poorer sleep quality.
Fatigue | 12 months
  Fatigue (as assessed by PROMIS-Fatigue Scale, Short Form 8 items): The NIH developed the Patient Reported Outcomes Measurement Information System (PROMIS®). The PROMIS Fatigue scale assesses a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The fatigue short forms are universal rather than disease-specific and assess fatigue over the past seven days (5 minutes).
The Trail Making Test (TMT) | 12 months
  The Trail Making Test (TMT) is one of the most popular neuropsychological tests and is included in most test batteries. The TMT provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions.
Verbal Fluency Test | 12 months
  The Verbal Fluency Test, consisting of the FAS, PRW, and CFL phonemic fluency subtests, will be administered across three distinct time points to reduce practice effects and to allow for a more reliable assessment of longitudinal change in executive function and lexical retrieval. Administering different letter sets at each visit minimizes familiarity with specific stimuli and provides a more valid evaluation of verbal generativity and cognitive flexibility over time.
Category Fluency Test | 12 months
  The Category Fluency Test, including the Animal Naming, Fruits and Vegetables Naming, and Cities and Towns Naming subtests, will be administered across three time points to assess semantic fluency while minimizing practice effects. Using a different semantic category at each visit reduces familiarity with specific item sets and provides a more accurate longitudinal measure of semantic memory retrieval, lexical access, and executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — University of California, Los Angeles